CLINICAL TRIAL: NCT03399565
Title: Children and Adolescent Registry for Diabetes Study in Jiangxi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, YunFeng Shen, professor, Second Affiliated Hospital of Nanchang University
Other Study IDs: SecondNanchangU
Record Dates: First submitted 2017-12-04; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to understand and evaluate different age children and adolescents with diabetes prevalence, self-management of disease , for diabetes patients and their families to provide diabetes management information, so as to help the children and adolescents diabetes patients to improve the quality of life.

DETAILED DESCRIPTION:
Background:With the development of economy and the improvement of people's living standards, the incidence of childhood diabetes is rapidly increasing.The multicenter, prospective,retrospectively in children and adolescents registry for diabetes in jiangxi aims to understand and evaluate different age children and adolescents with diabetes prevalence, self-management of disease , for diabetes patients and their families to provide diabetes management information, so as to help the children and adolescents diabetes patients to improve the quality of life.

Methods:The province's multi-center, prospective、retrospective study, the number of cases planned to be included in 300 cases.The inclusion criteria:A diagnosis of diabetes;reported for diabetes by parents and patients or by doctors and medical records to prove all of the patients;0-30 years old, gender not limited;voluntary participation and sign a consent form.Exclusion criteria

:At the same time, other test drugs or are other clinical trials;Due to other reasons, the researchers think that the person doesn't fit into the group;Diabetes during pregnancy;Besides diabetes diagnosis of tumor, cardiovascular disease and other interfere with the results of the study of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 days to 30 years who were diagnosed with diabetes according to the World Health Organization criteria;
* Gender is not limited.

Exclusion Criteria:

* Gestational diabetes mellitus;
* Patients with malignant tumor,cardiovascular disease and other interference with the results of the study of the disease.
* Patients are participating in any other clinical studies;

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Second Affiliated Hospital of Nanchang University
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01-18 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1C | About 3 months after the visit
  HbA1c <7%
blood pressure | About 3 months after the visit
  systolic blood pressure <130mm Hg, diastolic blood pressure<80mmHg
TC | About 3 months after the visit
  TC<5.2mmol/L
TG | About 3 months after the visit
  TG<1.7mmol/L
LDL-C | About 3 months after the visit
  LDL-C<2.6mmol/L
HDL-C | About 3 months after the visit
  HDL-C>1.0mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi, China